CLINICAL TRIAL: NCT06227520
Title: Acellular Dermal Allograft for Chronic Diabetic Wounds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-5933
Record Dates: First submitted 2024-01-10; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Wound Heal; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dermgen (Experimental): Application of Dermgen
  Interventions: Other: decellularized dermal matrix

INTERVENTIONS:
Other: decellularized dermal matrix — Application of Wound bed
  Other Names: Dermgen

SUMMARY:
The purpose of this study is to determine the efficacy of a novel decellularized dermal matrix (DDM) DermGEN™ for the treatment of diabetic foot ulcers (DFU). Despite several advances in wound treatments, hard-to-heal wounds, such as diabetic foot ulcer, still require 12 to 16 weeks to achieve complete closure. Although the focus of most research into wound-healing treatments has been on moisture and bacterial control, new approaches that target the instability of the extracellular matrix (ECM) in a wound are timely and much needed, particularly for hard-to-heal wounds such as DFUs. Innovative technologies that provide ECM interactions halt the chronic inflammatory cycle and stimulate cells that allow for tissue regeneration and wound healing. DermGEN™ is a human dermal allograft that has been minimally processed from human skin to remove epidermal and dermal cells while preserving the structure and intrinsic properties of the natural extracellular matrix of the dermis. This has potential to facilitate a shorter wound-healing time.

DETAILED DESCRIPTION:
DermGEN™ is a human dermal allograft that has been minimally processed from human skin to remove epidermal and dermal cells while preserving the structure and intrinsic properties of the natural extracellular matrix of the dermis. The resulting sterile decellularized scaffold provides a support for cellular repopulation and vascularization at the surgical site to facilitate integumental wound healing. Unlike other tissue-derived ECM-based products, such as acellular and decellularized matrices where treatments require anywhere from 6 to 10 reapplications of the product to achieve wound-closure rates of only 35% to 55% (16) DermGEN™ only requires one. A feasibility study has shown that 82% of participants (9 of 11 subjects) who had their DFU (1 ulcer/participant) treated with a single application of DDM (DermGEN) achieved complete wound closure between 2 and 8 weeks, with a mean 3.3 weeks and median of 2.3 weeks (https://doi.org/10.1016/j.jcjd.2022.03.010). The investigators have used this technology on a number of cases with good success. The investigators wish to gather further data with this study.

The purpose of this clinical trial is to perform a pilot study to determine the efficacy of DermGEN in the treatment in acute and non-healing diabetic foot ulcers (DFU). This will be a one-arm prospective study. It is hypothesized that DermGEN treatment will result in positive healing outcomes with no significant adverse effects. We anticipate to enroll 30 patients.

After enrolment and an initial assessment (time 0 data), participants will be treated with a single application of the DDM following standard-of-care procedures that include debridement of the DFU to provide healthy bleeding tissue margins. Then, it is applied with the dermal side in contact with the ulcer bed and covered by a bolster dressing. The bolster dressing is changed weekly during the follow-up. Follow-up assessments are conducted at 1, 2, 3, 4, 12 and 20 weeks. Digital photography is used to capture the appearance and size of the ulcer at each visit.

ELIGIBILITY:
Inclusion Criteria:

A subject will be considered eligible to participate in this study if each of the following inclusion criteria is satisfied:

1. Patient's ulcer has been present for a minimum of 2 weeks as of Day 0.
2. Study ulcer has healed <30% in size during the 2 weeks prior to Day 0.
3. Ulcer area is ≥1 cm2 prior to debridement at Day 0 of study.
4. Ulcer extends through dermis and into subcutaneous tissue but without exposure of muscle, tendon, bone or joint capsule.
5. Ulcer is free of necrotic debris and clinical infection, and is comprised of healthy vascular tissue suitable for skin grafting on Day 0.
6. Patient has adequate circulation to the foot as evidenced by toe pressure measurement.
7. Female patients are not pregnant at time of, or during study.
8. Patient and caregiver ready and willing to participate and comply with follow-up regime.
9. Patient or legal representative has read and signed the Institutional Ethics Review Board approved informed consent form.

Exclusion Criteria:

A subject will not be considered eligible to participate in this study if any one of the following exclusion criteria is satisfied:

1. Evidence of gangrene on affected foot.
2. Ulcer is over Charcot deformity (fractures or dislocation).
3. Ulcer is non-diabetic in etiology.
4. Patient receiving oral or parenteral corticosteroids, immunosuppression or cytotoxic agents, or is anticipated to require such agents during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 20 weeks
  Percentage of Wound Area Reduction Compared to Baseline

SECONDARY OUTCOMES:
Wound healing | 1 year
  Percentage of Patients with Complete Healing at Any Time Point
Adverse events | 20 weeks
  Number of Patients With Adverse Events
Ulcer Reoccurrence | 1 year
  Number of Patients with Ulcer Reoccurrence in the Same Location after Complete Healing

CONTACTS AND LOCATIONS:
Overall Officials: Graham Roche-Nagle, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costa IG, Glazebrook M, Lu S, McLaren AM, Gratzer PF. A Feasibility and Safety Study of a Novel Human Decellularized Dermal Matrix to Accelerate Healing of Neuropathic Diabetic Foot Ulcers in People With Type 1 and Type 2 Diabetes. Can J Diabetes. 2022 Oct;46(7):671-677. doi: 10.1016/j.jcjd.2022.03.010. Epub 2022 Apr 6. PMID 35945125